CLINICAL TRIAL: NCT00223158
Title: L-T3 Preparation for I131 Whole Body Scintigraphy: A Randomized Controlled Trial
Brief Title: Evaluation Study of L-T3 Utility in the Follow-up of Patients With Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrice Perron (Other)
Collaborators: Theramed co. (Unknown)
Responsible Party: Sponsor-Investigator, Patrice Perron, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRC 03-52-R1
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2005-07

CONDITIONS: Thyroid Cancer
Keywords: Thyroid cancer; Hypothyroidism; Whole Body Scintigraphy; Liothyronine; TSH elevation
MeSH Terms: conditions — Thyroid Neoplasms; Hypothyroidism | interventions — Triiodothyronine

INTERVENTIONS:
Drug: Liothyronine

SUMMARY:
To compare the hypothyroid state in patients with thyroid cancer prepared either by placebo or L-T3 following L-T4 withdrawal in preparation for whole body scintigraphy. To evaluate the time needed for TSH elevation (> 30 mUI/L) on placebo vs. L-T3.

DETAILED DESCRIPTION:
Patients with well differentiated thyroid cancer (DTC) need whole-body scintigraphy (WBS) and thyroglobulin (Tg) measurement in order to detect recurrence. Classically, withdrawal from levothyroxine (L-T4) during 4-6 weeks is needed for TSH elevation (> 30mUI/L), to allow iodine uptake and Tg production. As a result, patients become hypothyroid with impaired quality of life and a potential for tumour flare-up. Recombinant hTSH before WBS prevents hypothyroidism but is not yet approved for radioiodine treatment and is an expensive therapy. L-T3 substitution during the first 2-3 weeks of withdrawal is an alternative used empirically to prepare patients; however, no data exists to prove its benefit upon reducing hypothyroidism.

Objectives: 1) To compare the hypothyroid state in patients prepared either by placebo or L-T3 following L-T4 withdrawal. 2) To evaluate the time needed for TSH elevation (> 30 mUI/L) on placebo vs. L-T3.

Method: At the time of L-T4 withdrawal or after thyroidectomy, patients with DTC awaiting WBS or radioiodine treatment were randomized in two groups (double-blind): L-T3 (50 mg qd) or an identical placebo for 3 weeks, after which treatment was stopped for 2 weeks. A validated questionnaire of signs and symptoms of hypothyroidism (Billewicz's scale) was administered every 2 weeks until the WBS. TSH, fT4 and fT3 were measured weekly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with well-differentiated thyroid cancer, with total thyroidectomy
* 18 y.o. or older

Exclusion Criteria:

* Use of rhTSH for Whole Body Scintigraphy preparation
* Non stable cardiac arrythmias
* Any condition impairing TSH elevation(glucocorticoid use, hypopituitarism)
* Allergy to Liothyronine
* Inability to give a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2003-09; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the hypothyroid status by the Billewicz questionnaire.

SECONDARY OUTCOMES:
The time to reach an acceptable TSH elevation.

CONTACTS AND LOCATIONS:
Overall Officials: Rébecca Leboeuf, MD, Principal Investigator — Université de Sherbrooke; Marie-France Langlois, MD, Principal Investigator — Université de Sherbrooke; Patrice Perron, MD, Principal Investigator — Université de Sherbrooke; André Carpentier, MD, Principal Investigator — Université de Sherbrooke; Jean Verreault, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada